CLINICAL TRIAL: NCT02806362
Title: An Open-Label Study to Evaluate the Safety and Efficacy of Ombitasvir/Paritaprevir/Ritonavir in Japanese Adults With Genotype 1b Chronic Hepatitis C Virus (HCV) Infection With End Stage Renal Disease on Hemodialysis (GIFT-R)
Brief Title: Study of Ombitasvir/Paritaprevir/Ritonavir in Japanese Adults With Genotype 1b Chronic Hepatitis C Virus (HCV) Infection With End Stage Renal Disease (ESRD) on Hemodialysis (HD)
Acronym: GIFT-R
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-733
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Hepatitis C Virus
Keywords: Non-cirrhotic; End Stage Renal Disease (ESRD); moderate fibrosis; Chronic Hepatitis C Virus ( HCV); Chronic Hepatitis C Genotype 1b
MeSH Terms: conditions — Hepatitis C, Chronic; Kidney Failure, Chronic | interventions — ombitasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ombitasvir/paritaprevir/ritonavir (12 weeks) (Experimental): Ombitasvir/paritaprevir/ritonavir (25/50/100mg once daily) for 12 weeks
  Interventions: Drug: Ombitasvir/paritaprevir/ritonavir

INTERVENTIONS:
Drug: Ombitasvir/paritaprevir/ritonavir — Tablet

SUMMARY:
The purpose of this multicenter, single-arm, combination-drug study, which includes 12 weeks of treatment and 24 weeks of follow-up, is to evaluate the safety, efficacy and pharmacokinetics of ombitasvir/paritaprevir/ritonavir in Japanese adults infected with HCV GT1b, who are treatment-naïve or treatment-experienced to an IFN-based regimen and who have ESRD on HD.

ELIGIBILITY:
Inclusion Criteria:

* Females must be practicing specific forms of birth control on study treatment, or be post-menopausal for more than 2 years or surgically sterile
* Hepatitis C Virus (HCV) Ribonucleic acid (RNA) greater than 10,000 IU/mL at Screening
* Chronic HCV, Genotype (GT)1b infection
* Treatment-naive or treatment-experienced with an interferon (IFN)-containing regimen (IFN or pegylated-IFN with or without ribavirin).
* A fibrosis assessment test result equivalent to Metavir F0-F2.

Exclusion Criteria:

* Presence of Y93H variant at Screening
* Positive test result for Hepatitis B surface antigen (HBsAg) or anti-Human immunodeficiency virus antibody (HIV Ab)
* Significant liver disease with any cause other than chronic HCV infection
* On peritoneal dialysis
* On hemodialysis for more than 15 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2018-06 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving a 12-week sustained virologic response (SVR12). | 12 weeks after the last dose of study drug
  SVR12 defined as the hepatitis C virus (HCV) ribonucleic acid (RNA) level less than the lower limit of quantification (LLOQ) 12 weeks after the last dose of study drug.

SECONDARY OUTCOMES:
Percentage of participants with on-treatment virologic failure | Up to Week 12
  On-treatment virologic failure was defined as the following:
  Confirmed increase from nadir in HCV RNA (2 consecutive HCV RNA measurements greater than 1 log10 IU/mL above nadir) at any time point during treatment; or Confirmed HCV RNA greater than or equal to LLOQ after HCV RNA is less than LLOQ during treatment; or HCV RNA greater than or equal to LLOQ persistently during treatment with at least 6 weeks of treatment.
Percentage of participants with relapse | Up to 12 weeks after the last dose of study drug
  Participants with a confirmed HCV RNA greater than or equal to the LLOQ between Final treatment visit and 12 weeks after the last dose of study drug among participants completing treatment and with HCV RNA less than LLOQ at Final treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Koji Kato, MD, Study Director — AbbVie